CLINICAL TRIAL: NCT03860701
Title: Remote Ischemic Conditioning in Necrotizing Enterocolitis: Feasibility and Safety Pilot Study.
Brief Title: Remote Ischemic Conditioning in Necrotizing Enterocolitis
Status: Completed | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Agostino Pierro, Head of The Division of General and Thoracic Surgery, The Hospital for Sick Children
Other Study IDs: REB1000061144
Record Dates: First submitted 2019-01-17; First posted 2019-03-04 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Enterocolitis, Necrotizing
MeSH Terms: conditions — Enterocolitis, Necrotizing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Remote ischemic conditioning — An appropriately sized blood pressure cuff will be inflated around a limb (systolic blood pressure + 15 mmHg) for different periods of time (1 to up to 4 minutes), times (1 to up to 4 times) and consecutive days (1 to up to 2).

SUMMARY:
Necrotizing enterocolitis (NEC) affects up to 10% of very preterm infants. NEC mortality is high (30-50 %) and has remained unchanged over the last decades. New treatments are urgently needed. NEC pathogenesis is multifactorial, but bowel ischemia plays an essential role in NEC development. Remote ischemic conditioning (RIC) consists in inducing brief periods of non-lethal ischemia in a limb distant to an organ suffering from ischemia. RIC has been used in adults, children and term neonates with a variety of diagnosis. However, no study has been done including preterm infants with NEC.

DETAILED DESCRIPTION:
An appropriately sized blood pressure cuff will be applied to an arm or leg and inflated to promote RIC. This study will be conducted in three phases to assess the feasibility and safety of RIC in relation to duration of ischemia time, number of cycles of RIC and whether it is feasible and safe to perform RIC on consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NEC (stages I-III Bell's Classification)
* Weight greater or equal to 750 g.
* Gestational age < 36 weeks.
* Patients whose parents consent to participate in the study.

Exclusion Criteria:

* Patients with major congenital anomalies
* No antecedent of limb ischemia/limb thrombotic events.
* No antecedent diagnosis of occlusive arterial or venous thrombosis
* Hemodynamic instability

Ages: 0 Months to 3 Months | Sex: All
Age Groups: Child
Study Population: Preterm infants < 36 weeks with NEC (stages I-III as per Bell's modified classification).
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2018-12-17 (Actual); Primary Completion 2019-08-20 (Actual); Study Completion 2019-08-20 (Actual)

PRIMARY OUTCOMES:
Limb perfusion after Remote Ischemic Conditioning | 1 days
  Limb perfusion will be assessed before (baseline) and after Remote Ischemic Conditioning (RIC). Limb perfusion will be determined by oxygen saturation using pulse oximetry. RIC will be considered feasible and safe if the procedure is completed as planned with no failure of limb re-perfusion. Failure is defined as no return of limb arterial oxygen saturation to baseline 4 minutes after the ischemic phase (re-perfusion time).

SECONDARY OUTCOMES:
Cutaneous injury | 1 days
  Defined as new-onset skin breakdown, bruising, ecchymosis or petechiae.
Persistent pain | 1 days
  Pain measured according to the premature infant pain profile (PIPP) scores (range 0-21). Pain scores will be obtained immediately before (baseline) and 6 hours after RIC. Persistent pain will be defined as a PIPP score higher than the baseline score.

CONTACTS AND LOCATIONS:
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zozaya C, Ganji N, Li B, Janssen Lok M, Lee C, Koike Y, Gauda E, Offringa M, Eaton S, Shah PS, Pierro A. Remote ischaemic conditioning in necrotising enterocolitis: a phase I feasibility and safety study. Arch Dis Child Fetal Neonatal Ed. 2023 Jan;108(1):69-76. doi: 10.1136/archdischild-2022-324174. Epub 2022 Aug 8. PMID 35940871